CLINICAL TRIAL: NCT03958799
Title: Safety and Immunogenicity of an Investigational Tetanus Toxoid, Reduced Diphtheria Toxoid, and Acellular Pertussis Adsorbed (Tdap) Vaccine in Young Adults
Brief Title: A Study to Describe the Safety Profile and Compare the Immune Response of 4 Different Formulations of an Investigational Tdap Vaccine When Compared to Licensed Tdap Vaccine in Young Adults in Canada
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NGB00005; U1111-1217-2612 (Other: UTN)
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Tetanus Immunisation (Healthy Volunteers); Diphtheria Immunisation (Healthy Volunteers); Pertussis Immunisation (Healthy Volunteers)

STUDY DESIGN:
Intervention Model Description: Modified double-blind: the study participant, the Investigator, and other study personnel remain unaware of the treatment assignments throughout the trial. An unblinded vaccine administrator will administer the appropriate vaccine but will not be involved in safety assessment and data collection.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Group 1: Investigational Product (IP) Formulation A (Experimental): IP Formulation A administration, participation in Stage 1 and Stage 2
  Interventions: Biological: Investigational Tdap vaccine Formulation A
- Group 2: IP Formulation A (Experimental): IP Formulation A administration, participation in Stage 1
  Interventions: Biological: Investigational Tdap vaccine Formulation A
- Group 3: IP Formulation B (Experimental): IP Formulation B administration, participation in Stage 1 and Stage 2
  Interventions: Biological: Investigational Tdap vaccine Formulation B
- Group 4: IP Formulation B (Experimental): IP Formulation B administration, participation in Stage 1
  Interventions: Biological: Investigational Tdap vaccine Formulation B
- Group 5: IP Formulation C (Experimental): IP Formulation C administration, participation in Stage 1 and Stage 2
  Interventions: Biological: Investigational Tdap vaccine Formulation C
- Group 6: IP Formulation C (Experimental): IP Formulation C administration, participation in Stage 1 and Stage 2
  Interventions: Biological: Investigational Tdap vaccine Formulation C
- Group 7: IP Formulation D (Experimental): IP Formulation D administration, participation in Stage 1 and Stage 2
  Interventions: Biological: Investigational Tdap vaccine Formulation D
- Group 8: Tdap (Active Comparator): TdaP administration, participation in Stage 1 and Stage 2
  Interventions: Biological: Licensed Tdap vaccine
- Group 9: Tdap (Active Comparator): TdaP administration, participation in Stage 1
  Interventions: Biological: Licensed Tdap vaccine

INTERVENTIONS:
Biological: Investigational Tdap vaccine Formulation B — Pharmaceutical form:Suspension for injection Route of administration: Intramuscular
  Arms: Group 3: IP Formulation B; Group 4: IP Formulation B
Biological: Investigational Tdap vaccine Formulation C — Pharmaceutical form:Suspension for injection Route of administration: Intramuscular
  Arms: Group 5: IP Formulation C; Group 6: IP Formulation C
Biological: Investigational Tdap vaccine Formulation A — Pharmaceutical form:Suspension for injection Route of administration: Intramuscular
  Arms: Group 1: Investigational Product (IP) Formulation A; Group 2: IP Formulation A
Biological: Investigational Tdap vaccine Formulation D — Pharmaceutical form:Suspension for injection Route of administration: Intramuscular
  Arms: Group 7: IP Formulation D
Biological: Licensed Tdap vaccine — Pharmaceutical form:Suspension for injection Route of administration: Intramuscular
  Arms: Group 8: Tdap; Group 9: Tdap

SUMMARY:
The primary objectives of this study are:

* To describe the safety profile of each of the investigational vaccine formulations for all participants
* To describe the humoral and cell-mediated immune responses to all of the investigational vaccine formulations
* To evaluate the dose response to vaccine components
* To describe the magnitude, quality, and longevity of immune responses to each of the investigational vaccine formulations

DETAILED DESCRIPTION:
Study duration per participant is approximately 1 year, which will include a safety follow-up contact at 12 months after vaccination

ELIGIBILITY:
Inclusion criteria :

* Individuals born in Canada and vaccinated with a combination vaccine in accordance with the National Immunization Program (NIP).
* Aged ≥ 19 years and < 22 years on the day of inclusion.
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion criteria:

* Pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 3 months after the last vaccination. To be considered of non-childbearing potential, a female must be pre-menarche, or post-menopausal for at least 1 year, or surgically sterile.
* Participation at the time of study enrollment (or in the 4 weeks preceding the first trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine in the 4 weeks before and/or after any study vaccination except for influenza vaccination only, which may be received at least 2 weeks before or 2 weeks after any study vaccination.
* History of autoimmune disorder.
* History of cardiovascular disorder.
* History of Guillain-Barré syndrome.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances.
* Laboratory-confirmed/self-reported thrombocytopenia, contraindicating intramuscular vaccination.
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0 C). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 19 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting immediate adverse events (AEs) | Within 30 minutes post-vaccination
  AEs, including those related to the product administered
Number of participants reporting solicited injection sites or systemic reactions | Within 7 days post-vaccination
  Solicited reaction: adverse reaction prelisted in the case report book (CRB) Injection site reactions: pain, erythema, swelling Systemic reactions: fever, headache, malaise, myalgia, arthralgia, chills
Number of participants reporting unsolicited AEs | Within 30 days post-vaccination
  AEs other than solicited reactions
Number of participants reporting serious adverse events (SAEs) | Up to 12 months post-vaccination
  SAEs, including adverse event of special interest (AESIs)
Number of participants reporting medically attended adverse events (MAAEs) | Up to 12 months post-vaccination
  MAAE: a new onset or a worsening of a condition that prompts the participant to seek unplanned medical advice at a physician's office or emergency department
Number of participants reporting adverse events of special interest (AESIs) | Up to 12 months post-vaccination
  AESIs are reported until the end of the safety follow-up period
Number of participants reporting Grade 2 and Grade 3 laboratory parameter abnormalities | Within 60 days post-vaccination
  Haematological and biochemical laboratory parameters
Geometric mean concentrations (GMCs) of anti-pertussis antigen immunoglobulins | From Day 0 to Day 360
  Anti-pertussis antigen immunoglobulins concentration will be measured by mesoscale discovery electrochemiluminescence (MSD ECL)
GMCs of anti-diphtheria toxoid immunoglobulins | From Day 0 to Day 360
  Anti-diphtheria toxoid total immunoglobulins concentration will be measured by MSD ECL
GMCs of anti-tetanus toxoid immunoglobulins | From Day 0 to Day 360
  Anti-tetanus toxoid total immunoglobulins concentration will be measured by MSD ECL
Geometric means of antigen-specific cells | From Day 0 to Day 360
  Antigen specific cells will be measured by FLUOROSPOT
Percentages of antigen-specific cells | From Day 0 to Day 360
  Antigen specific cells will be measured by FLUOROSPOT

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (5):
- Canada (5):
  - Investigational Site Number 1240006, Halifax
  - Investigational Site Number 1240009, Pierrefonds
  - Investigational Site Number 1240004, Québec
  - Investigational Site Number 1240005, Sherbrooke
  - Investigational Site Number 1240003, Truro

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org